CLINICAL TRIAL: NCT04643028
Title: Comparison of Effectiveness of Mulligan Mobilization Technique and Cervical Stabilization Training in Patients With Chronic Neck Pain: A Single-Blinded Randomized Controlled Trial
Brief Title: Effectiveness of Mulligan Mobilization Technique And Cervical Stabilization Training in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Serbay SEKEROZ (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Serbay SEKEROZ, Research Assistant, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/53905
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator who made the outcome measurements will not have any information about the group of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home exercise (Other): The exercise program will include active normal joint movements in the cervical region, postural exercises, strengthening exercises for the scapular retractor muscles, and stretching exercises for the pectoral muscles, levator scapula and upper part of the trapezius and breathing/relaxation exercises.
  Interventions: Other: Home exercise
- Mulligan mobilization (Other): Mulligan mobilization will be applied to this group in addition to the exercises in the home exercise group. In painless directions, each session will be applied in 3 sets, a set of 10 repetitions. Sixty seconds of rest will be given between sets.
  Interventions: Other: Mulligan mobilization
- Cervical stabilization (Other): In addition to the exercises in the home exercise group, this group will be given cervical stabilization training that focuses on the deep neck muscles.
  Interventions: Other: Cervical stabilization

INTERVENTIONS:
Other: Home exercise — Exercise program will include active normal joint movements in the cervical region, postural exercises, strengthening exercises for the scapular retractor muscles, and stretching exercises for the pectoral muscles, levator scapula and upper part of the trapezius and breathing/relaxation exercises.
  Arms: Home exercise
Other: Mulligan mobilization — Mulligan mobilization: Mulligan mobilization will be applied to this group in addition to the exercises in the home exercise group. In painless directions, each session will be applied in 3 sets, a set of 10 repetitions.Sixty seconds of rest will be given between sets.
  Arms: Mulligan mobilization
Other: Cervical stabilization — Cervical stabilization group: In addition to the exercises in the home exercise group, this group will be given cervical stabilization training that focuses on the deep neck muscles.
  Arms: Cervical stabilization

SUMMARY:
The aim of our study is to compare the efficiency of Mulligan mobilization technique and cervical stabilization training in patients with chronic neck pain. The results obtained from the study will contribute to the planning of the treatment of patients with chronic neck pain more effectively.

DETAILED DESCRIPTION:
The aim of our study is to compare the efficiency of Mulligan mobilization technique and cervical stabilization training in patients with chronic neck pain. The results obtained from the study will contribute to the planning of the treatment of patients with chronic neck pain more effectively.

The hypotheses we will test for this purpose; H1. Home exercise program will improve positively after treatment in patients with chronic neck pain compared to before treatment.

H2. Mulligan mobilization will improve positively after treatment in patients with chronic neck pain compared to before treatment.

H3. Cervical stabilization training will improve positively after treatment in patients with chronic neck pain compared to before treatment.

H4. Mulligan mobilization will provide more effective results in patients with chronic neck pain compared to other applications.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain lasting more than 3 months
* Expressing neck pain at least 3,5/10 points and above on a Visual Analog Scale
* Being 18-65 years old
* Agree to participate in the study
* Having obtained 5/50 points and above in Neck Disability Index

Exclusion Criteria:

* Having had spinal surgery
* Other musculoskeletal problems that may affect the cervical region such as impingement, thoracic outlet and scoliosis.
* Having a diagnosed psychiatric illness
* Having benefited from physiotherapy and / or another treatment method due to spinal pain problem in the last 1 year.
* The presence of specific pathological conditions such as malignant condition, fracture, systemic rheumatoid disease.
* Any health problem that may prevent the application of evaluations and / or treatment other than those mentioned above.
* Difficulty in communication at a level that prevents the application of evaluations and / or treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 5 minutes
  Pain intensity will be evaluated with the Visual Analogue Scale. The Visual Analogue Scale is a horizontal scale in the range of 0-10 cm, where 0 is the lowest pain and 10 the highest pain. The patient will be asked to mark the pain felt in the neck area on this line and the point marked will be measured with a ruler and recorded in cm.
Neck Disability | 5 minutes
  Neck Disability will be measured by Neck Disability Index. The Neck Disability Index is a frequently used scale to evaluate the level of disability due to neck pain. It consists of 10 items and 6 options under each item. Options are scored between 0-5 points. An increasing score indicates a higher level of disability.
Cervical Range of Motion | 5 minutes
  Cervical Range of Motion will be assessed by Baseline Bubble Inclinometer as degree of flexion-extension, rotation and lateral flexion and will be recorded.
Head Posture | 5 minutes
  Head posture will be evaluated using the craniovertebral angle. The decrease in the craniovertebral angle indicates an increased anterior head posture.
Proprioception | 5 minutes
  The "joint position sense error test" defined by Revel et al. Will be used to evaluate cervical proprioception.
Muscle Endurance | 3 minutes
  "Cervical Deep Flexor Muscle Endurance Test" will be used.
Neck Awareness | 5 minutes
  The Fremantle Neck Awareness Questionnaire, which consists of few and short questions, does not take time, is easy to access, evaluates neck perception, attention and proprioceptive awareness, will be used. An increase in the score obtained from the questionnaire indicates a decrease in neck awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Aslan Telci, Professor, Study Director — Professor